CLINICAL TRIAL: NCT04840160
Title: Influence of Tart Cherry Juice Intervention on Vascular Function and the Urinary Metabolite; a Preliminary Study to Inform Study Design
Brief Title: Influence of Tart Cherry Juice Intervention on Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: lucymurray2016
Record Dates: First submitted 2021-04-06; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Dietary Exposure; Metabolic Disturbance
Keywords: cherry; anthocyanin; vascular function; metabolomics

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Investigator
Masking Description: Participants supplied with treatment or placebo in a plastic container
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants supplied with 30 ml of a low fruit (<1%) cordial mixed with maltodextrin and protein diluted in 100 ml water twice daily, once in the morning and evening.
  Interventions: Dietary Supplement: Placebo
- Cherry juice (Experimental): Participants supplied with 30 ml of a tart cherry juice concentrate (CherryActive, United Kingdom; (containing 36.8 mg of anthocyanins) diluted in 100 ml of water twice daily, once in the morning and evening.
  Interventions: Dietary Supplement: Cherry juice

INTERVENTIONS:
Dietary Supplement: Cherry juice — A tart cherry juice intervention
  Arms: Cherry juice
Dietary Supplement: Placebo — A tart cherry juice placebo
  Arms: Placebo

SUMMARY:
Diets containing fruit rich in anthocyanins have been shown (in meta-analyses) to be beneficial for health, but intervention trials have shown inconsistent results. In this preliminary study we want to investigate the influence of a tart-cherry juice intervention on vascular function and explore metabolite profiles that may offer insight into their mechanism of action

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the primary cause of morbidity and mortality. Tart cherries (TC) can positively impact major risk factors of CVD, activities thought to be related to their phytochemical content. However, data from human trials is less clear. TC have been shown to reduce systolic blood pressure (SBP) after acute, short-term and chronic intake, and to improve vascular dysfunction, presumably due to their antioxidant and anti-inflammatory activities. Other studies have not shown benefits of TC on SBP or vascular function and studies are difficult to interpret with different populations, dosing and durations being used as well as a lack of understanding for any underlying mechanisms. To account for the latter, the use of metabolomics has become increasingly popular in nutritional research. Therefore, the aim of this preliminary study was to characterise the effects of TC supplementation on vascular function with a 4-week intervention and explore if metabolomics can provide mechanistic evidence and this will inform for future chronic studies with TC juice.

ELIGIBILITY:
Inclusion Criteria:

* aged 19-40
* no diagnosed issues with the ability to consume fruit juice
* no known food intolerances to fruits

Exclusion Criteria:

* participants that are cigarette smokers
* participants diagnosed with hypertension
* participants diagnosed with any form of cardiometabolic diseases
* participants that require any prescribed prescriptions excluding the contraceptive pill
* participants that are regular consumers of cherries (>100 g/d)
* participants that consume any antioxidant supplements

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressure | Change in blood pressure following 4 weeks intervention
  Measurement of systolic and diastolic blood pressure before and after the intervention
Arterial pulse wave velocity | Change in pulse wave velocity following 4 weeks intervention
  Measurement of pulse wave velocity before and after the intervention
Digital volume pulse | Change in digital volume pulse following 4 weeks intervention
  Measurement of digital volume pulse before and after the intervention

SECONDARY OUTCOMES:
Metabolomics | Changes to urinary metabolite profiles following 4 weeks intervention
  Ion intensities of ca 5000 metabolites in urine samples before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Glyn Howatson, Principal Investigator — Northumbria University
Locations (1):
- Northumberland Building, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Research data will be shared on request